CLINICAL TRIAL: NCT03394716
Title: Monitoring MRI Changes Before and During Radiotherapy Treatment of Brain Tumors
Status: Terminated | Type: Observational
Why Stopped: Low inclusion rate; Change of position of principal investigator.
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: N17MRB
Record Dates: First submitted 2017-11-28; First posted 2018-01-09 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Brain Tumor
Keywords: MRI; Radiotherapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient brain tumor treated with fractionated radiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — standard radiotherapy treatment with 1-3 extra MRIs

SUMMARY:
This study aims to evaluate anatomical and functional changes during RT for patients receiving fractionated RT for brain tumors. Anatomical changes during RT will be registered and analyzed and if needed the radiotherapy plan will be modified for the individual patient. This means that the "to be irradiated volume" will be modified according to the shape changes of the tumor. The functional MRI sequences will be used to evaluate what parameters, and at which time point, are important for radiotherapy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Primary brain tumor (WHO IV, GBM); treated with fractionated radiotherapy with or without preceding surgery. Systemic treatment is allowed before and during radiotherapy.
* Brain metastasis (from a solid extracranial tumor) eligible for treatment with fractionated radiotherapy with or without preceding surgery. Systemic treatment is allowed before and during radiotherapy.

Also, postoperative patients with a macroscopic residual tumor lesion can be included (the diagnosis of residual diseases is defined by the treating neurosurgeon or on the MRI executed within 24 hours after the surgery, the diagnosis of residual macroscopic disease should always be confirmed during the neuro-oncology multidisciplinary meeting).

Exclusion Criteria:

* Patients receiving Whole Brain RT (WBRT)
* Patient with a poor kidney function (GFR < 30 mL/min; CKD 4 and 5; patients on dialysis and patients with acute kidney insufficiency)
* None, doubtful or very small (<5 mm in its largest dimension) contrast enhancing lesion
* Patients with a contraindication for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastasis in the brain from extracranial solid tumors or patients with primary brain tumors who will be treated with fractionated radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
MRI parameters in the target volume | through study completion, an average of 3 years
  functional MRI parameters (permeability, perfusion and diffusion) in the target volume before and during fractional radiotherapy treatment
anatomical variations in position, shape and size in the target volume | through study completion, an average of 3 years
  The difference is position shape and size in the target volume before and during fractional radiotherapy treatment. In case there is no macroscopic extension beyond the clinical target volume the new target volumes (gross target volume (GTV) and clinical target volume (CTV).) will also (but later) be delineated for analysis of volume changes, center of mass changes and distance measurements between the delineation on planning MRI versus repeated MRI.

SECONDARY OUTCOMES:
the correlation between MRI parameters to the treatment outcome | through study completion, an average of 3 years
  to make a sample size calculation for a future study of imaging marker discovery.
the correlation between anatomical variations and the treatment outcome | through study completion, an average of 3 years
  to make a sample size calculation for a future study of imaging marker discovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No